CLINICAL TRIAL: NCT05270356
Title: MINDS Imaging Ancillary Study
Acronym: MINDS
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Boston Children's Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Rafael Ceschin, Assistant Professor, University of Pittsburgh
Other Study IDs: STUDY21020073; R01HL152740 (NIH)
Record Dates: First submitted 2022-02-01; First posted 2022-03-08 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2024-12

CONDITIONS: Adult Congenital Heart Disease
Keywords: Adult Congenital Heart Disease; Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MRI — Magnet Resonance Imaging of the Brain without Contrast

SUMMARY:
This study is an ancillary study to the NHLBI-funded Pediatric Heart Network (PHN) "Multi-Institutional Neurocognitive Discovery Study" (MINDS) in Adult Congenital Heart Disease (ACHD). The MINDS-ACHD" study will recruit 500 complex CHD patients between18-30 years old. The investigators propose to quantitate multi-modal neuroimaging biomarkers (brain injury, structure and physiology) which are not only important components of brain and cognitive reserve but can be predictive of neurocognitive decline and early onset of dementia in the aging non-CHD population.

DETAILED DESCRIPTION:
Dramatic advances in management of congenital heart disease (CHD) have improved survival to adulthood from <10% in the 1960's to nearly 90% in the current era. With this shifting demographic, adult CHD (ACHD) patients now outnumber pediatric CHD patients. ACHD patients demonstrate domain-specific neurocognitive deficits such as impairment in executive function, associated with reduced quality of life that includes deficits in educational attainment and social interaction. These deficits are related to risk factors that can occur across the lifespan, including genetic abnormalities, cumulative hypoxic/ischemic injury, and, adult-onset atherosclerotic cerebrovascular disease. The overarching hypothesis is that ACHD patients exhibit vascular brain injury and structural/physiological brain alterations that are predictive of specific neurocognitive deficits, including executive dysfunction, which are modified by behavioral and environmental enrichment proxies of CR (e.g., level of education and lifestyle/social habits). The investigators propose an ancillary study to the NHLBI-funded Pediatric Heart Network (PHN) "Multi-Institutional Neurocognitive Discovery Study (MINDS) in Adult Congenital Heart Disease (ACHD)." The investigators will leverage the MINDS-ACHD parent study data (i.e., NIH Toolbox neuropsychological battery/clinical data/biological samples) and an established neuroimaging harmonization, which the investigators currently use for the PHN Single Ventricle Reconstruction (SVRIII) multi-center brain connectome study (R01-HL128818), to measure neuroimaging biomarkers in ACHD patients at the same PHN sites. The specific aims are: Specific Aim #1 (brain injury): To determine if vascular-related brain injury (cortical infarcts, hemosiderin lesions, and white matter hyperintensity) is associated with specific neurocognitive deficits (e.g. NIH Toolbox total composite score) in ACHD patients. Specific Aim #2 (brain structure): To determine if reduced fronto-temporal cortical thickness and white matter connectivity are associated with specific neurocognitive deficits (e.g. NIH Toolbox frontal executive sub-score) in ACHD patients. Specific Aim #3 (brain physiology): To determine if reduced cerebrovascular reserve (regional cerebral blood flow/ resting BOLD imaging) is associated with specific neurocognitive deficits (e.g. NIH Toolbox crystallized composite score) in ACHD patients. Specific Aim #4 (cognitive reserve): To determine if the associations between neuroimaging biomarkers and neurocognitive outcomes in ACHD patients are modified by behavioral and environmental enrichment proxies of CR, using traditional statistical models and machine learning techniques. Given the paucity of multi-modal neuroimaging studies in ACHD, the proposed study addresses a major knowledge gap in the ACHD population by providing insight into the mechanism underlying impaired neurocognitive outcomes. This study will provide structural-physiological correlates of neurocognitive outcomes, representing the first multi-center neuroimaging study to be performed in ACHD. Importantly, other behavioral and environmental enrichment data will be integrated with these neuroimaging and neurocognitive outcome data to model cognitive reserve. Results from this research will help shape the care of ACHD patients, and further our understanding of the interplay between brain injury and cognitive reserve. The proposed ancillary study is thus both feasible and cost-effective by leveraging the NHLBI-PHN infrastructure. As such, the proposed research is well aligned with the NHLBI's Strategic Vision.

ELIGIBILITY:
Inclusion Criteria:

• Participation in and completion of MINDS parent study procedures. The inclusion criteria for the MINDS parent study consists of ACHD patients aged 18 - 30 years with moderate and severely complex CHD.

Exclusion Criteria:

* Individuals with mild complexity lesions;
* Individuals with MRI contraindications will be excluded from study participation. Contraindications include, but are not limited, to:
* Pregnancy or breast feeding
* Claustrophobia or inability to lie still for an extended period
* Implantable device (i.e., pacemaker; defibrillator; ferromagnetic aneurysm clips; cochlear implant; gastric reflux device; internal insulin pump; pacing leads; neurostimulation system) that cannot be cleared for scanning at 3T
* Foreign body (i.e., metallic splinter in the eye; bullet or grenade fragments)
* Braces or orthodontic appliances that cannot be removed prior to scanning and/or cannot be cleared for scanning at 3T
* Individuals who are unable to participate in the informed consent process or complete the study questionnaire will also be excluded from participation.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Males and Females aged 18 to 30 who have been diagnosed with Congenital Heart Disease
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Brain Injury | At time of MRI
  Vascular-related brain injury (cortical infarcts, hemosiderin lesions, and white matter hyperintensity)

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Panigrahy, MD, Principal Investigator — University of Pittsburgh
Locations (13):
- United States (12):
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cohen S, Earing MG. Neurocognitive Impairment and Its Long-term Impact on Adults With Congenital Heart Disease. Prog Cardiovasc Dis. 2018 Sep-Oct;61(3-4):287-293. doi: 10.1016/j.pcad.2018.08.002. Epub 2018 Aug 15. PMID 30118722
- [Background] Daliento L, Mapelli D, Russo G, Scarso P, Limongi F, Iannizzi P, Melendugno A, Mazzotti E, Volpe B. Health related quality of life in adults with repaired tetralogy of Fallot: psychosocial and cognitive outcomes. Heart. 2005 Feb;91(2):213-8. doi: 10.1136/hrt.2003.029280. PMID 15657236
- [Background] Utens EM, Bieman HJ, Verhulst FC, Meijboom FJ, Erdman RA, Hess J. Psychopathology in young adults with congenital heart disease. Follow-up results. Eur Heart J. 1998 Apr;19(4):647-51. doi: 10.1053/euhj.1997.0824. PMID 9597415
- [Background] Utens EM, Verhulst FC, Erdman RA, Meijboom FJ, Duivenvoorden HJ, Bos E, Roelandt JR, Hess J. Psychosocial functioning of young adults after surgical correction for congenital heart disease in childhood: a follow-up study. J Psychosom Res. 1994 Oct;38(7):745-58. doi: 10.1016/0022-3999(94)90027-2. PMID 7877129
- [Background] Ilardi D, Ono KE, McCartney R, Book W, Stringer AY. Neurocognitive functioning in adults with congenital heart disease. Congenit Heart Dis. 2017 Mar;12(2):166-173. doi: 10.1111/chd.12434. Epub 2016 Dec 13. PMID 27957813
- [Background] Murphy LK, Compas BE, Reeslund KL, Gindville MC, Mah ML, Markham LW, Jordan LC. Cognitive and attentional functioning in adolescents and young adults with Tetralogy of Fallot and d-transposition of the great arteries. Child Neuropsychol. 2017 Jan;23(1):99-110. doi: 10.1080/09297049.2015.1087488. Epub 2015 Sep 20. PMID 26388325
- [Background] Klouda L, Franklin WJ, Saraf A, Parekh DR, Schwartz DD. Neurocognitive and executive functioning in adult survivors of congenital heart disease. Congenit Heart Dis. 2017 Jan;12(1):91-98. doi: 10.1111/chd.12409. Epub 2016 Sep 21. PMID 27650247